CLINICAL TRIAL: NCT04049227
Title: A Pilot, Multicenter, Single Arm, Open Label, Surgical Window of Opportunity Study of Abemaciclib and Letrozole for Endometrioid Adenocarcinoma of the Endometrium
Brief Title: Abemaciclib and Letrozole in Treating Patients With Endometrial Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 18G07; STU00209370 (CTRP (Clinical Trial Reporting Program)); NU 18G07 (Other: Northwestern University); P30CA060553 (NIH); NCI-2019-04599 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-07-31; First posted 2019-08-08 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Endometrial Endometrioid Adenocarcinoma
MeSH Terms: interventions — abemaciclib; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (letrozole, abemaciclib) (Experimental): Patients receive letrozole PO QD and abemaciclib PO BID on days 1-14. Patients then undergo standard of care hysterectomy on day 15.
  Interventions: Drug: Abemaciclib; Drug: Letrozole; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Abemaciclib — Given PO
  Other Names: LY-2835219; LY2835219; Verzenio
Drug: Letrozole — Given PO
  Other Names: CGS 20267; Femara
Procedure: Therapeutic Conventional Surgery — Undergo standard of care hysterectomy

SUMMARY:
This early phase I trial studies how well abemaciclib and letrozole work in treating patients with endometrial cancer and determines whether there are changes in patients' cancer cell biomarkers (a genetic feature or specific protein) for cell growth before and after treatment. Antihormone therapy with aromatase inhibitors, such as letrozole, may lessen the amount of estrogen made by the body. Abemaciclib blocks the activities of a class of proteins called cyclin-dependent kinase, which are involved in cell duplication. Giving letrozole and abemaciclib together may slow down cancer cell growth in patients with endometrial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether there are changes in Ki-67 expression from the pretreatment specimen (e.g. biopsy or dilation and curettage [D&C]) to the post-treatment hysterectomy specimen following treatment with letrozole and abemaciclib.

SECONDARY OBJECTIVES:

I. To determine the proportion of tumors with complete cell cycle arrest (CCCA) response as measured by Ki-67 expression between the pre-treatment tumor and the posttreatment tumor.

II. To identify biological characteristics of tumors (e.g. mismatch repair [MMR] status, PTEN mutational status, etc.) correlating with decreased Ki-67 expression induced by the letrozole and abemaciclib combination.

III. To determine the frequency of adverse events associated with use of abemaciclib and letrozole.

EXPLORATORY OBJECTIVES:

I. To evaluate the correlation of the expression of Ki-67 with that of cyclin D1, p16, pRB, and PTEN as well as with MMR deficiency.

OUTLINE:

Patients receive letrozole orally (PO) once daily (QD) and abemaciclib PO twice daily (BID) on days 1-14. Patients then undergo standard of care hysterectomy on day 15.

After completion of study treatment, patients are followed up at 30 days and at 2 and 6 weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a new histologically confirmed diagnosis of endometrioid adenocarcinoma of the endometrium who are candidates for hysterectomy.

  * Note: Patients with recurrent disease are not eligible.
* Patients must be willing to provide archival tumor biopsy slides from the specimen (e.g. endometrial biopsy or dilation and curettage) which diagnosed them with endometrial cancer.

  * (Please note: Given the amount of tissue obtained from these specimens is often much more than a core needle biopsy, we do not anticipate difficulties with insufficient tissue.)
* Patients should be treatment naive. They should not have received any endometrial cancer directed therapy including medroxyprogesterone acetate, aromatase inhibitors, other hormonal treatments or radiation therapy for treatment of endometrial cancer.

  * Note: Patients can have used oral contraceptives or hormonal replacement therapy provided these were discontinued 28 days prior to trial enrollment.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 within 28 days prior to registration for protocol therapy.
* Patients must have adequate organ function for all of the following criteria within 28 days of registration.
* Absolute neutrophil count (ANC) >= 1.5 x 10^9 /L (within 28 days of registration).
* Platelets >= 100 x 10^9 /L (within 28 days of registration).
* Hemoglobin >= 8 g/dL (within 28 days of registration).

  * Patients may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin earlier than the day after the erythrocyte transfusion.
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (within 28 days of registration).

  * Patients with Gilbert?s syndrome with a total bilirubin =< 2.0 times ULN and direct bilirubin within normal limits are permitted.
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN (within 28 days of registration).
* Serum creatinine =< 1.5 x ULN (within 28 days of registration).
* Patients with a history of surgical sterilization are eligible for this study. OR
* Patients must have post-menopausal status due to menopause (surgical or natural). Patients must meet at least one of the following criteria:

  * Bilateral oophorectomy
  * Age >= 55 years
  * Age =< 55 years and amenorrhea (absence of menstruation) for > 12 months OR
* Patients who are not post-menopausal or previously sterilized.

  * i.e. a female of childbearing potential (patients who are not post-menopausal), must have a negative serum pregnancy test within 7 days of the first dose of study treatment (abemaciclib and/or letrozole). Patient must agree to use adequate birth control (condoms with spermicidal agent or abstinence) while on the study and for 3 weeks after completion of treatment.
* Patients should be able to swallow oral medications.
* Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study.
* Patients must be willing and able to have a window of >= 15 days prior to their scheduled hysterectomy surgery after registration.

Exclusion Criteria:

* Patients who have had chemotherapy, hormonal therapy or radiotherapy directed at the treatment of endometrial cancer prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks prior to registration are not eligible.
* Patients may not be receiving any other investigational agents. A wash out period of 4 weeks before registration is required for eligibility.
* Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to abemaciclib or letrozole or any of its excipients are not eligible.
* Patients receiving CYP3A inducers or strong CYP3A inhibitors will not be eligible for this study. A wash-out period of minimum 5 half-lives or 7 days, whichever is shorter, before registration is required for the patient to become eligible.
* Patients who have a known personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest are not eligible.
* Patients who have known active bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus [HIV] positivity or with known active hepatitis B or C (for example, hepatitis B surface antigen positive). Screening is not required for enrollment.

  * Note: patients with uncomplicated urinary tract infection or uncomplicated cystitis are eligible.
* Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following, are not eligible:

  * Hypertension that is not controlled on medication
  * Baseline grade 2 or higher diarrhea.
  * Ongoing or active infection requiring systemic treatment.
  * Symptomatic congestive heart failure.
  * Unstable angina pectoris.
  * Psychiatric illness that would limit compliance with study requirements.
  * Social situations that would limit compliance with study requirements.
  * Serious preexisting medical condition(s) that would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, history of major surgical resection involving the stomach or small bowel, or preexisting Crohn?s disease or ulcerative colitis or a preexisting chronic condition resulting in baseline grade 2 or higher diarrhea).
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient?s safety or study endpoints.
* Female patients who are pregnant or nursing are not eligible.
* Patients who are unable to retain oral medication, and patients who have gastrointestinal disorders or abnormalities that would interfere with absorption of the study drugs are not eligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Changes in Ki-67 expression | Baseline up to 6 weeks

SECONDARY OUTCOMES:
Proportion of tumors with complete cell cycle arrest (CCCA) response | At day 15
  Will be measured by Ki-67 between the pre-treatment tumor and the post-treatment tumor. CCCA response is defined as less than 3% of tumor cells staining positive for Ki-67 from specimens obtained at time of hysterectomy. Baseline biomarker levels will be compared between patients who do vs.
  do not achieve complete CCCA using a two-sample t-test.
Biological characteristics of tumors: MMR status | Up to 6 weeks
  Will be measured to correlate with decreased Ki-67 expression induced by the letrozole and abemaciclib combination.
Biological characteristics of tumors: PTEN mutational status | Up to 6 weeks
  Will be measured to correlate with decreased Ki-67 expression induced by the letrozole and abemaciclib combination.
Biological characteristics of tumors: expression of cyclin D1 | Up to 6 weeks
  Will be measured to correlate with decreased Ki-67 expression induced by the letrozole and abemaciclib combination.
Biological characteristics of tumors: p16 | Up to 6 weeks
  Will be measured to correlate with decreased Ki-67 expression induced by the letrozole and abemaciclib combination.
Biological characteristics of tumors: pRB | Up to 6 weeks
  Will be measured to correlate with decreased Ki-67 expression induced by the letrozole and abemaciclib combination.
Incidence of adverse events associated with abemaciclib and letrozole | Up to 6 weeks
  Categorized and graded according to Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Barber, MD, MS, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois